CLINICAL TRIAL: NCT01693900
Title: Efficacy of Fascia Iliaca Block Versus Intraoperative Nerve Infiltration During Anterior Hip Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Randy Fayne, DO (Other)
Responsible Party: Sponsor-Investigator, Randy Fayne, DO, Principle Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-285
Record Dates: First submitted 2012-08-23; First posted 2012-09-26 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2017-08

CONDITIONS: Pain, Postoperative
Keywords: joint replacement; total hip replacement; regional pain block; ultrasound guidance; fascia iliaca compartment block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-operative Ultrasound FICB Group (Experimental): Enrolled subjects will receive FICB with 50cc of 0.3% ropivacaine. Blocks will be performed under an ultrasound guidance device with an in-plane technique by a single study investigator, in the preoperative area.
  Interventions: Procedure: Pre-operative Ultrasound FICB Group
- Intra-operative FICB Group (Active Comparator): Enrolled subjects will receive FICB with 50cc of 0.3% ropivacaine. Blocks will be performed intra-operatively under direct surgeon visualization, in the operating room.
  Interventions: Procedure: Intra-operative FICB Group

INTERVENTIONS:
Procedure: Pre-operative Ultrasound FICB Group — Enrolled subjects will receive FICB with 50cc of 0.3% ropivacaine. Blocks will be performed under ultrasound guidance with an in-plane technique by a single study investigator in the preoperative area. Although possible without ultrasound guidance, using this technique allows for identification of specific tissue planes and precise placement of medication near the nerves responsible for postoperative pain. Using ultrasound, the superficial fascial layer of the iliopsoas muscle is identified at the anterior edge of the ilium, and a needle is placed just beneath that fascia. A high volume of local anesthetic is then injected under ultrasound guidance, ensuring cephalad spread of medication in an attempt to provide anesthesia of the lateral femoral cutaneous, femoral and obturator nerves.
  Arms: Pre-operative Ultrasound FICB Group
Procedure: Intra-operative FICB Group — Enrolled subjects will receive FICB with 50cc of 0.3% ropivacaine. Blocks will be performed intra-operatively under direct surgeon visualization, in the operating room. Unlike other approaches to hip replacement, anterior repair allows for direct visualization of the fascial layers described above. This allows for direct injection of local anesthetic beneath this fascia, potentially obviating the need for preoperatively performed, ultrasound guided, FICB.
  Arms: Intra-operative FICB Group

SUMMARY:
Surgical trauma causes nerve sensitization leading to amplification and prolongation of postoperative pain. In experimental studies, pre-injury neural blockade using local anesthetics has been shown to reduce post-injury sensitization of the central nervous system, while similar techniques applied after the injury had less or no effect (FILOS). Investigators have therefore designed this study to examine the timing of FICB (pre-operatively versus intra-operatively) on postoperative pain in patients undergoing anterior hip replacement surgery.

DETAILED DESCRIPTION:
Though still uncommonly used in the United States, the popularity of the anterior approach for total hip replacement is rapidly growing because of its clinical advantages. Rehabilitation is simplified and accelerated, dislocation risk is reduced, leg length is more accurately controlled, and incision is smaller than with traditional approaches (GOEBEL). Nevertheless, although pain is lessened, it is still considerable, and new techniques have been developed to improve postoperative pain control for this procedure.

Surgical incision and tissue trauma result in postoperative pain. Regional pain blocks, especially when done under ultrasound guidance, have proven to be extremely effective at reducing postoperative pain and improving patient satisfaction. One such block, the fascia iliaca compartment block (FICB), has been shown to be effective in controlling pain associated with surgery involving the hip and femur.

Although possible without ultrasound guidance, using this technique allows for identification of specific tissue planes and precise placement of medication near the nerves responsible for postoperative pain. Using ultrasound, the superficial fascial layer of the iliopsoas muscle is identified at the anterior edge of the ilium, and a needle is placed just beneath that fascia. A high volume of local anesthetic is then injected under ultrasound guidance, ensuring cephalad spread of medication, in an attempt to provide anesthesia of the lateral femoral cutaneous, femoral and obturator nerves.

Unlike other approaches to hip replacement, anterior repair allows for direct visualization of the fascial layers described above. This allows for direct injection of local anesthetic beneath this fascia, potentially obviating the need for preoperatively performed, ultrasound guided, FICB. The primary differences in approach (ultrasound guided preop versus direct visualization intraop) is the timing of injection, and it is unclear if nerve block prior to or after tissue damage affects postoperative pain in these patients.

Surgical trauma causes nerve sensitization leading to amplification and prolongation of postoperative pain. In experimental studies, pre-injury neural blockade using local anesthetics has been shown to reduce post-injury sensitization of the central nervous system, while similar techniques applied after the injury had less or no effect (FILOS). Investigators have therefore designed this study to examine the timing of FICB (pre-operatively versus intra-operatively) on postoperative pain in patients undergoing anterior hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* Female patients must be surgically sterile, postmenopausal or have a negative pregnancy test on the day of surgery
* Willing and able to sign the informed consent approved by the Institutional Review Board (IRB)
* Willing and able to complete the study procedures and pain scales, and to communicate meaningfully in English with study personnel
* Elective anterior hip replacement to be performed at Beaumont Hospital, Royal Oak
* American Society of Anesthesiologists physical status classification 1, 2, and 3 (patients that have either no systemic illness, or mild to moderate systemic disease, eg. asthma, diabetes or hypertension)

Exclusion Criteria:

* History of allergy to study medications including ropivacaine and other local anesthetic agents of the amide-type
* Enrollment in concurrent research study
* Female patients who are pregnant or lactating, or who have a positive urine pregnancy test
* Opioid tolerant, ie, A patient taking a narcotic > 30mg per day morphine equivalent. (Source: www.globalrph.com/narcotic.cgi) for pain in the 2 months prior to surgery
* A medical condition that in the investigator's opinion could adversely impact the patient's participation or safety, conducts of the study, or interferes with the pain assessments
* Previous hip arthroplasty (partial or total) of the index hip
* History of illicit drug use, or prescription medicine or alcohol abuse within the past 2 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randy Fayne, DO, Principal Investigator — Beaumont Health
Locations (1):
- Beaumont Health System, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-center, prospective, randomized study enrolled 50 subjects who were scheduled for elective anterior hip replacement. Once informed consent was obtained, patients were randomized to either preoperative ultrasound-guided fascia iliaca compartment block (FICB) or intraoperative surgeon-placed FICB.
Groups:
- Pre-operative Ultrasound FICB Group: Enrolled subjects will receive FICB with 50cc of 0.3% ropivacaine. Blocks will be performed under an ultrasound guidance device with an in-plane technique by a single study investigator, in the preoperative area.
  Pre-operative Ultrasound FICB Group: 25 subjects will receive FICB with 50cc of 0.3% ropivacaine. Blocks will be performed under an ultrasound guidance device with an in-plane technique by a single study investigator, in the preoperative area.
- Intra-operative FICB Group: Enrolled subjects will receive FICB with 50cc of 0.3% ropivacaine. Blocks will be performed intra-operatively under direct surgeon visualization, in the operating room.
  Intra-operative FICB Group: 25 subjects will receive FICB with 50cc of 0.3% ropivacaine. Blocks will be performed intra-operatively under direct surgeon visualization, in the operating room. Unlike other approaches to hip replacement, anterior repair allows for direct visualization of the fascial layers described above. This allows for direct injection of local anesthetic beneath this fascia, potentially obviating the need for preoperatively performed, ultrasound guided, FICB.
Period: Overall Study
Arm/Group | Pre-operative Ultrasound FICB Group | Intra-operative FICB Group
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data lost for one participant in Intra-operative FICB group leaving 24 analyzed for all measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-operative Ultrasound FICB Group | Intra-operative FICB Group | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 10 | 12 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain During PACU Admission
Description: Pain assessments will be made by the subject using a 10.0 cm Visual-Analog scale (VAS) (scale 1-100 where 1=minimal pain and 100= worst pain imaginable) as follows at each time point:
  * Baseline assessment in Preoperative area
  * Upon arrival to the post-anesthesia care unit (PACU)
  * Every 15 min (+/- 2 minutes) thereafter and prior to any request for pain medication until PACU discharge All pain scores per subject from the time of PACU admission until discharge from PACU will be averaged to obtain one data point per subject.
Time Frame: From time of PACU admission until discharge from PACU, an average of 2 hours
Population: Data lost for one participant in Intra-operative FICB group leaving 24 analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pre-operative Ultrasound FICB Group | Intra-operative FICB Group
Number analyzed (Participants) | 25 | 24
units on a scale | 40 [35 to 44] | 36 [26 to 47]

2. Primary Outcome: Postoperative Pain During Recovery
Description: Pain assessments were made by the subject using a 10.0 cm VAS (scale 1-100 where 1=minimal pain and 100= worst pain imaginable) prior to any request for pain medication. Up to 40 values per patient were averaged.
Time Frame: From discharge from PACU until discharge from hospital, an average of 2-3 days
Population: Data not available for 1 patient in Pre-operative ultrasound FICB group and 3 patients Intra-operative FICB group
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pre-operative Ultrasound FICB Group | Intra-operative FICB Group
Number analyzed (Participants) | 24 | 22
units on a scale | 25 [15 to 50] | 26 [11 to 38]

3. Secondary Outcome: Incidence of Adverse Events
Description: Measure is count of participants experiencing any adverse event. Adverse events will be reported by the patient (or when appropriate, staff personnel) during hospitalization.
Time Frame: From the signature on the informed consent document for the duration of the hospital stay, an expected average of 2 - 3 days.
Population: Data lost for one participant in Intra-operative FICB group leaving 24 analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Ultrasound FICB Group | Intra-operative FICB Group
Number analyzed (Participants) | 25 | 24
Participants | 20 | 19

4. Secondary Outcome: Patient Satisfaction With Postoperative Pain Control
Description: Patient satisfaction with postoperative pain control, using a 10 point Likert scale where 1=extremely dissatisfied and 10= extremely satisfied. Patients were called 3 weeks post-op to determine pain control satisfaction.
Time Frame: At the 3 week post-op visit
Population: Data was obtained for the 25 patients in the pre-operative group and 22 patients in the intra-operative group who responded to 3-week followup phone calls.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pre-operative Ultrasound FICB Group | Intra-operative FICB Group
Number analyzed (Participants) | 25 | 22
units on a scale | 9.7 (0.6) | 8.8 (2.2)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from time of consent until end of study at the 3 week-postoperative assessment.
Arm/Group | Pre-operative Ultrasound FICB Group | Intra-operative FICB Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 6/25 | 11/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-operative Ultrasound FICB Group (N=25) | Intra-operative FICB Group (N=24)
Dizziness (General disorders) | 1 (1) | 1 (1)
Shivering (General disorders) | 1 (1) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Swelling of knee/thigh (General disorders) | 0 (0) | 1 (1)
Swelling of lips (General disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute blood loss anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Tape burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size limited conclusions that could be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No